CLINICAL TRIAL: NCT02872428
Title: A Phase 1, Single Ascending Dose, Double Blind, Placebo Controlled Study to Evaluate the Safety and Tolerability of Valproic Acid in Healthy Volunteers (Part 1) or Trauma Patients(Part 2)
Brief Title: A Study to Evaluate the Safety and Tolerability of Valproic Acid in Trauma Patients(Part 2)
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: at request of funding group because of failure to enroll more than one patient
Sponsor: Dr. Hasan Alam (Other)
Responsible Party: Sponsor-Investigator, Dr. Hasan Alam, Hasan Alam, MD, Norman Thompson Professor of Surgery Section Head, General Surgery, University of Michigan
Organization: University of Michigan (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: HUM00067452; VPA-C-002 (Other Grant/Funding Number: Department of Defense/ONR)
Record Dates: First submitted 2016-05-23; First posted 2016-08-19 (Estimated); Last update posted 2017-11-06 (Actual); Status verified 2017-10

CONDITIONS: Shock,Hemorrhagic; Trauma
MeSH Terms: conditions — Shock, Hemorrhagic; Wounds and Injuries | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Valproic acid (Depacon) (Experimental): Valproic acid by IV infusion over one hour
  Interventions: Drug: Valproic Acid
- Isotonic saline solution (Placebo Comparator): The placebo administered by IV infusion over 1 hour
  Interventions: Drug: Isotonic saline solution

INTERVENTIONS:
Drug: Valproic Acid — By infusion over 1 hour
  Other Names: Depacon
  Arms: Valproic acid (Depacon)
Drug: Isotonic saline solution — By infusion over 1 hour
  Arms: Isotonic saline solution

SUMMARY:
THIS IS THE SECOND PART OF A 2-PART STUDY. The purpose of the first part of this study was to determine the safety and tolerability of ascending doses of valproic acid (also known as Depacon) administered as intravenous infusion (IV) in doses ranging from 15 mg/kg to 250 mg/kg in healthy subjects.

ID: VPA-C-002

The second part of the study will also be to determine the safety and tolerability of single ascending doses of valproic acid administered as IV in trauma subjects with hemorrhagic shock.

DETAILED DESCRIPTION:
THIS IS THE SECOND PART OF A 2-PART STUDY. Part 1 of the study will be a single center study intended to assess the safety and tolerability of valproic acid dosages at 15 mg/kg, 30 mg/kg, 60 mg/kg, 90 mg/kg, 120 mg/kg, 150 mg/kg 180 mg/kg, 210 mg/kg and 250 mg/kg. Up to 72 healthy subjects (9 dose groups of 8 subjects) will receive single doses of valproic acid or placebo via a 60-min IV infusion in a ratio of 3:1 active drug: placebo. ID: VPA-C-002

Part 2 of the study will be a multi-center, double blind, placebo-controlled study in trauma patients with hemorrhagic shock. The patients will be able to consent themselves, or if unable due to injuries, a Legally Authorized Representative will consent for them. Up to 12 patients (2 dose groups of 6 patients) will receive single doses of valproic acid or placebo via a 60-min IV infusion in a ratio of 2:1 active drug : placebo. The dose levels in Part 2 will be the two highest doses that are demonstrated to have acceptable safety profile based on the review of safety data from Part 1 (130mg/kg and 140mg/kg).

ELIGIBILITY:
Inclusion Criteria:

1. Male and non-pregnant female trauma patients between the ages of 18-70 years, inclusive.
2. Blunt or penetrating trauma resulting in two or more systolic blood pressure readings of ≤ 110 mmHg at any point during transport to the hospital or within the first hour after arrival in the emergency department. Systolic blood pressure readings of ≤ 110 mmHg need not be consecutive (Eastridge et al., 2007).
3. Patient's admission to the emergency department results in trauma team activation (per institutional criteria, see Appendix 7).
4. Patient's injuries are considered potentially survivable by the attending trauma surgeon on initial evaluation.
5. Able to provide informed consent or consent can be obtained from a representative (spouse or other legally authorized representative) in the event that the subject is unconscious or otherwise impaired.
6. Female subjects must be postmenopausal, surgically sterilized, or have a negative urinary pregnancy test on arrival. Criteria for menopause include age > 45 with absence of menses for > 12 months. Criteria for surgical sterilization include hysterectomy and/or oophorectomy. Tubal ligation with menses within the past 12 months is not considered to be surgical sterilization.
7. Body mass index (BMI) between 18 kg/m2 and 35 kg/m2

Exclusion Criteria:

1. Subjects with known history of adverse reaction to Valproic acid.
2. Subjects with known history of hepatitis B or C or clinical history of hepatic dysfunction, pancreatitis, or renal insufficiency.
3. Subjects with -amylase >400 U/L or lipase >300 U/L or creatinine >ULN
4. Subjects with AST or ALT >3X Upper limit of normal (ULN) or total bilirubin >1.5X Upper limit of normal (ULN)
5. Subjects with 2nd or 3rd degree burns of any size and location.
6. Female subjects who are pregnant or lactating.
7. Subjects who are currently incarcerated.
8. Subjects with severe traumatic brain injury (with Glasgow Coma Scale score <8 on arrival to the emergency department).
9. Non-hemorrhagic causes of shock, including septic, cardiogenic, or neurogenic shock or mechanical reasons such as tension pneumothorax or cardiac temponade.
10. Subjects with inadequate venous access.
11. Subject with a hemoglobin level of less than 8g/dL.

    -

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-09-29 (Actual); Study Completion 2017-09-29 (Actual)

PRIMARY OUTCOMES:
Dose limiting toxicity (DLT) | As this is a safety study, subjects will be monitored for side-effects beginning immediately after the one hour infusion until the follow-up visit (between 2-6 weeks post infusion) is completed.
  Dose limiting toxicity (DLT) will be measured by drug-related grade 2 (moderate) or higher
  toxicity indicators (excluding fever, chills, nausea or other possible infusion-related effects).

CONTACTS AND LOCATIONS:
Overall Officials: Hasan Alam, MD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - The University of Michigan, Ann Arbor, Michigan